CLINICAL TRIAL: NCT03859960
Title: The Effects of Spasticity on Glucose Metabolism and Soft Tissue Body Composition in Individuals With Motor Complete and Motor Incomplete Spinal Cord Injury
Brief Title: The Effects of Spasticity on Glucose Metabolism in Individuals With Spinal Cord Injury
Status: Completed | Type: Observational
Sponsor: Fatih Sultan Mehmet Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Arzu Atici, Principal Investigator, Fatih Sultan Mehmet Training and Research Hospital
Other Study IDs: 2013/22
Record Dates: First submitted 2019-02-26; First posted 2019-03-01 (Actual); Results first posted 2020-09-04 (Actual); Last update posted 2020-09-04 (Actual); Status verified 2020-08

CONDITIONS: Spinal Cord Injuries
Keywords: Body composition; glucose; spasticity; spinal cord injury
MeSH Terms: conditions — Spinal Cord Injuries; Muscle Spasticity | interventions — Body Composition; Absorptiometry, Photon

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: body composition — fat mass % (FM%) and fat-free mass (FFM%)% of arms, legs, trunk, android, gynoid and total body
  Other Names: dual-energy absorptiometry (DXA),
Diagnostic Test: glucose, insulin, glycohemoglobin — In the morning after 12 hours overnight fast, all individuals underwent a 75 gram (g) oral glucose tolerance test (OGTT). Blood samples were taken before loading glucose and then 30, 60, 90 and 120 minutes after taking glucose solution in order to measure serum glucose and insulin levels. Glycohemoglobin (HbA1c) was measured in blood samples taken before the OGTT. We calculated the Matsuda index and Homeostasis model assessment index (HOMA-IR) using glucose and insulin levels.
  Other Names: fasting blood glucose, insulin, glycohemoglobin

SUMMARY:
Muscle atrophy may occur in individuals with spinal cord injury (SCI) as a result of diminished physical activity and alterations in glucose metabolism and body composition may be seen. In a few studies, it has been suggested that spasticity may have a positive impact on glucose metabolism by preventing muscle atrophy and alterations in body composition in individuals with motor complete SCI. Investigators aimed to assess the effects of spasticity on glucose metabolism and body composition in participants with complete and incomplete SCI.

DETAILED DESCRIPTION:
Investigators plan a prospective clinical trial. Participants with SCI were included to study if times from injury were at least one year. Participants had an AIS grades of A-D with spasticity. We evaluated that participants with AIS A and B SCI were motor complete group, AIS C and D SCI were motor incomplete group. Spasticity was assessed with Modified Ashworth Scale (MAS) and spasms were assessed with Penn Spasm Frequency Scale (PSFS). Hip adductor and extensor spasticity, knee extensor and flexor spasticity and ankle plantar flexor spasticity were assessed by using MAS. Body composition was measured by dual-energy x-ray absorptiometry. All participants underwent a 75 gram (g) oral glucose tolerance test (OGTT). Insulin sensitivity was assessed by calculating Matsuda index and HOMA-IR. Investigators assessed the effects of spasticity on glucose metabolism and body composition in participants with SCI.

ELIGIBILITY:
Inclusion Criteria:

• Spinal cord injury AIS A,B,C,D

Exclusion Criteria:

* Other central nervous system diseases
* Significant complications that affect spasticity
* Joint contracture
* Diabetes mellitus

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals with SCI were included to study if they were 18-65 years old and times from injury were at least one year.
Sampling Method: Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2014-09-21 (Actual); Primary Completion 2018-05-10 (Actual); Study Completion 2018-08-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arzu Atici, Principal Investigator — Fatih Sultan Mehmet Training and Research Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Skold C, Levi R, Seiger A. Spasticity after traumatic spinal cord injury: nature, severity, and location. Arch Phys Med Rehabil. 1999 Dec;80(12):1548-57. doi: 10.1016/s0003-9993(99)90329-5. PMID 10597805
- [Background] Gorgey AS, Dudley GA. Spasticity may defend skeletal muscle size and composition after incomplete spinal cord injury. Spinal Cord. 2008 Feb;46(2):96-102. doi: 10.1038/sj.sc.3102087. Epub 2007 Jul 17. PMID 17637764
- [Background] Gorgey AS, Dolbow DR, Dolbow JD, Khalil RK, Castillo C, Gater DR. Effects of spinal cord injury on body composition and metabolic profile - part I. J Spinal Cord Med. 2014 Nov;37(6):693-702. doi: 10.1179/2045772314Y.0000000245. Epub 2014 Jul 7. PMID 25001559
- [Background] Gorgey AS, Dudley GA. Skeletal muscle atrophy and increased intramuscular fat after incomplete spinal cord injury. Spinal Cord. 2007 Apr;45(4):304-9. doi: 10.1038/sj.sc.3101968. Epub 2006 Aug 29. PMID 16940987
- [Background] Gorgey AS, Chiodo AE, Zemper ED, Hornyak JE, Rodriguez GM, Gater DR. Relationship of spasticity to soft tissue body composition and the metabolic profile in persons with chronic motor complete spinal cord injury. J Spinal Cord Med. 2010;33(1):6-15. doi: 10.1080/10790268.2010.11689669. PMID 20397439
- [Background] Jung IY, Kim HR, Chun SM, Leigh JH, Shin HI. Severe spasticity in lower extremities is associated with reduced adiposity and lower fasting plasma glucose level in persons with spinal cord injury. Spinal Cord. 2017 Apr;55(4):378-382. doi: 10.1038/sc.2016.132. Epub 2016 Sep 13. PMID 27618974

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Individuals with SCI recruited from the inpatient rehabilitation unit of an education and research hospital. Recruitment began in September 2014 and was completed in May 2018.
Groups:
- Motor Complete Group: Individuals with American Spinal Injury Association (ASIA) Impairment Scale grades A and B.
- Motor Incomplete Group: Individuals with American Spinal Injury Association (ASIA) Impairment Scale grades C and D.
Period: Overall Study
Arm/Group | Motor Complete Group | Motor Incomplete Group
Started | 14 | 19
Completed | 14 | 19
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: ASIA impairment scale (AIS) is the most prominent standardized clinical grading and classification method for the assessment of patients with spinal cord injury (SCI). Patients with AIS A and B are motor complete group, AIS C and D are motor incomplete group.
Groups:
- Motor Complete Group: Individuals with American Spinal Injury Association Impairment Scale (AIS) grades A and B.
- Motor Incomplete Group: Individuals with American Spinal Injury Association Impairment Scale (AIS) grades C and D.
- Total: Total of all reporting groups
Arm/Group | Motor Complete Group | Motor Incomplete Group | Total
Number analyzed (Participants) | 14 | 19 | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 19 | 33
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 4 | 11
  Male | 7 | 15 | 22
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 14 | 19 | 33
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Turkey | 14 | 19 | 33
Time since injury [Mean (Standard Deviation); unit: months] | 47.4 (52.6) | 62.1 (47.8) | 55.85 (49.63)

OUTCOME MEASURES:

1. Primary Outcome: Correlation Between Knee Flexor Muscle Modified Ashworth Scale and Insulin Resistance
Description: Modified Ashworth Scale is used to assess muscle spasticity on a 6-point scale. 0: No increase in muscle tone 4: Affected part(s) is (are) rigid in flexion or extension. Higher scores mean a worse outcome. HOMA index was used to evaluate insulin resistance. HOMA index is a simple, and inexpensive method used for evaluating insulin sensitivity. In most of the studies, values >2.7 were accepted as insulin resistance. HOMA-IR was calculated by using fasting plasma glucose (mg/dL) X fasting insulin (uIU/mL) /405 formula. Pearson correlation was used to calculate the correlation coefficient (r).
Time Frame: One day
Population: Individuals with spinal cord injury AIS A and AIS B (motor complete) and AIS C and D (motor incomplete) were evaluated. These 2 groups were not compared to each other. Each 2 groups were evaluated separately.
Measure: Number; unit: correlation coefficient
Groups:
- Motor Complete: American Spinal Injury Association Impairment Scale (AIS) Grades of A, B
- Motor Incomplete: American Spinal Injury Association Impairment Scale (AIS) Grades of C, D
Arm/Group | Motor Complete | Motor Incomplete
Number analyzed (Participants) | 14 | 19
correlation coefficient | -0.692 | 0.23
Statistical Analysis 1: Comparison: Motor Complete; Test type: Other; p = 0.006, Pearson correlation test
Statistical Analysis 2: Comparison: Motor Incomplete; Test type: Other; p = 0.23, Pearson correlation test — p<0.05 was considered statisticaly significant

2. Primary Outcome: Correlation Between Knee Flexor Muscle Modified Ashworth Scale and Insulin Sensitivity
Description: We used the Matsuda index to assess insulin sensitivity. Matsuda index was calculated 10.000/square root (Fasting plasma glucose x fasting plasma insulin) x (mean OGTT glucose concentration X mean OGTT insulin concentration) formula. Higher scores mean better. Modified Ashworth Scale is used to assess muscle spasticity on a 6-point scale. 0: No increase in muscle tone 4: Affected part(s) is (are) rigid in flexion or extension. Higher scores mean a worse outcome. Pearson correlation was used to calculate the correlation coefficient (r).
Time Frame: One day
Population: as for outcome 1
Measure: Number; unit: correlation coefficient
Arm/Group | Motor Complete | Motor Incomplete
Number analyzed (Participants) | 14 | 19
correlation coefficient | 0.797 | -0.084
Statistical Analysis 1: Comparison: Motor Complete; Test type: Other; p = 0.001, Pearson correlation test — p<0.05 was considered statisticaly significant
Statistical Analysis 2: Comparison: Motor Incomplete; Test type: Other; p = 0.731, Pearson correlation test

3. Primary Outcome: Correlation Between Penn Spasm Frequency Scale and Insulin Resistance
Description: Penn Spasm Frequency Scale is used to assess spasms. This scale is a 5-point scale. Higher scores mean a worse outcome. HOMA index is a simple, and inexpensive method used for evaluating insulin sensitivity. In most of the studies, values >2.7 were accepted as insulin resistance. HOMA-IR was calculated by using fasting plasma glucose (mg/dL) X fasting insulin (uIU/mL) /405 formula. Pearson correlation was used to calculate the correlation coefficient (r).
Time Frame: One day
Population: as for outcome 1
Measure: Number; unit: correlation coefficient
Groups:
- Motor Complete Group: Individuals with American Spinal Injury Association Impairment Scale (AIS) grade A and B.
Arm/Group | Motor Complete Group | Motor Incomplete Group
Number analyzed (Participants) | 14 | 19
correlation coefficient | 0.354 | -0.002
Statistical Analysis 1: Comparison: Motor Complete Group; Test type: Other; p = 0.214, Pearson correlation test
Statistical Analysis 2: Comparison: Motor Incomplete Group; Test type: Other; p = 0.993, Pearson correlation test — p<0.05 was considered statisticaly significant

4. Primary Outcome: Correlation Between Penn Spasm Frequency Scale and Insulin Sensitivity
Description: We used the Matsuda index to assess insulin sensitivity. Matsuda index was calculated 10.000/square root (Fasting plasma glucose x fasting plasma insulin) x (mean OGTT glucose concentration X mean OGTT insulin concentration) formula. Higher scores mean better. Penn Spasm Frequency Scale is used to assess spasms. This scale is a 5-point scale. Higher scores mean a worse outcome. Pearson correlation was used to calculate the correlation coefficient (r).
Time Frame: One day
Population: as for outcome 1
Measure: Number; unit: correlation coefficient
Arm/Group | Motor Complete | Motor Incomplete
Number analyzed (Participants) | 14 | 19
correlation coefficient | 0.289 | -0.103
Statistical Analysis 1: Comparison: Motor Complete; Test type: Other; p = 0.41, Pearson correlation test
Statistical Analysis 2: Comparison: Motor Incomplete; Test type: Other; p = 0.676, Pearson correlation test

5. Primary Outcome: Correlation Between Knee Flexor Muscle Modified Ashworth Scale and Total Body Fat-Free Mass%
Description: The body composition of the individuals was measured by dual-energy absorptiometry (DXA) device. Modified Ashworth Scale is used to assess muscle spasticity on a 6-point scale. 0: No increase in muscle tone 4: Affected part(s) is (are) rigid in flexion or extension. Higher scores mean a worse outcome. Pearson correlation was used to calculate correlation coefficient.
Time Frame: One day
Population: as for outcome 1
Measure: Number; unit: correlation coefficient
Arm/Group | Motor Complete | Motor Incomplete
Number analyzed (Participants) | 14 | 19
correlation coefficient | 0.201 | 0.287
Statistical Analysis 1: Comparison: Motor Complete; Test type: Other; p = 0.511, Pearson correlation test — p<0.05 was considered statisticaly significant
Statistical Analysis 2: Comparison: Motor Incomplete; Test type: Other; p = 0.248, Pearson correlation test

6. Primary Outcome: Correlation Between Penn Spasm Frequency Scale and Total Body Fat-Free Mass%
Description: The body composition of the individuals was measured by dual-energy absorptiometry (DXA) device. Penn Spasm Frequency Scale is used to assess spasms. This scale is a 5-point scale. Higher scores mean a worse outcome. Pearson correlation was used to calculate the correlation coefficient (r).
Time Frame: One day
Measure: Number; unit: correlation coefficient
Arm/Group | Motor Complete | Motor Incomplete
Number analyzed (Participants) | 14 | 19
correlation coefficient | -0.138 | 0.526
Statistical Analysis 1: Comparison: Motor Complete; Test type: Other; p = 0.654, Pearson correlation test
Statistical Analysis 2: Comparison: Motor Incomplete; Test type: Other; p = 0.025, Pearson correlation test

ADVERSE EVENTS:
Time Frame: One day
Groups:
- Motor Complete: individuals with AIS A, B
- Motor Incomplete: individuals with AIS C, D
Arm/Group | Motor Complete | Motor Incomplete
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/19
Other Adverse Events (participants affected / at risk) | 0/14 | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2020-08-06): https://cdn.clinicaltrials.gov/large-docs/60/NCT03859960/Prot_000.pdf
  • Statistical Analysis Plan (2020-08-06): https://cdn.clinicaltrials.gov/large-docs/60/NCT03859960/SAP_001.pdf
  • Informed Consent Form (2020-08-06): https://cdn.clinicaltrials.gov/large-docs/60/NCT03859960/ICF_002.pdf